CLINICAL TRIAL: NCT01550744
Title: A Phase 3b, Randomized, Double-blind, Active-controlled, Multicenter Study to Evaluate a "Subject-tailored" Maintenance Dosing Approach in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Study of Ustekinumab to Evaluate a "Subject-tailored" Maintenance Dosing Approach in Subjects With Moderate-to-Severe Plaque Psoriasis
Acronym: PSTELLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR100708; CNTO1275PSO3009 (Other: Janssen Biotech, Inc)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Psoriasis
Keywords: Psoriasis; Ustekinumab; STELARA; Skin disease; Monoclonal
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Approved q12w maintenance regimen (Experimental): Active ustekinumab study agent q12 weeks with sham/placebo as necessary to maintain blind
  Interventions: Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg; Drug: Placebo
- Group 2: Subject-tailored fixed-interval maintenance regimen (Experimental): Subjects will undergo placebo withdrawal and will receive active study agent up to q24w intervals with sham/placebo injections to maintain the blind.
  Interventions: Drug: Ustekinumab 45 mg; Drug: Ustekinumab 90 mg; Drug: Placebo

INTERVENTIONS:
Drug: Ustekinumab 45 mg — Form = Injection, route = subcutaneous
Drug: Ustekinumab 90 mg — Form = Injection, route = subcutaneous
Drug: Placebo — Form = Injection, route = subcutaneous

SUMMARY:
The purpose of the study is to assess the effect of extending maintenance dosing intervals beyond 12 weeks on the clinical efficacy and safety of ustekinumab in subjects with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
In this study, a proportion of subjects will receive study agent at its recommended dose and interval (45mg for subjects less than or equal to 100kg, or 90mg for subjects greater than 100kg; every 12 weeks after 2 starter doses at Weeks 0 and 4). The majority of subjects will have the opportunity to receive study agent less frequently during the randomization period depending on the subject's response. The study consists of a 4-week screening period; a 28-week open-label run-in period; a double-blind treatment period from Week 28 to Week 104; a 12 week post-treatment period; and a 20-week safety follow-up. Participants will be randomized for the double blind period into one of two study groups. Group 1 participants will receive an injection of the study medication at a 12 week dosing interval. Group 2 participants will undergo a placebo withdrawal and may receive study agents at an extended interval greater than 12 weeks. During the double-blind treatment period, subjects in Groups 1 and 2 will receive placebo as necessary to maintain the blind.

ELIGIBILITY:
Key Eligibility Criteria

* Male or female
* Have had a diagnosis of plaque-type psoriasis at least 6 months prior to the first administration of study agent (subjects with concurrent psoriatic arthritis may be enrolled).
* Have plaque-type psoriasis covering at least 10% of their total BSA at screening and at the time of the first administration of study agent.
* Have a PGA score of ≥ 3 at screening and at the time of the first administration of study agent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech, Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.
Locations (40):
- United States (40):
  - Birmingham, Alabama
  - Bakersfield, California
  - Irvine, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Santa Monica, California
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Coral Gables, Florida
  - Saint Augustine, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Plainfield, Indiana
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Troy, Michigan
  - Fridley, Minnesota
  - St Louis, Missouri
  - Henderson, Nevada
  - Lebanon, New Hampshire
  - East Windsor, New Jersey
  - New York, New York
  - The Bronx, New York
  - Williamsville, New York
  - Gahanna, Ohio
  - Norman, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Yardley, Pennsylvania
  - Johnston, Rhode Island
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Spokane, Washington
  - Clarksburg, West Virginia

REFERENCES:
- [Derived] Loesche MA, Farahi K, Capone K, Fakharzadeh S, Blauvelt A, Duffin KC, DePrimo SE, Munoz-Elias EJ, Brodmerkel C, Dasgupta B, Chevrier M, Smith K, Horwinski J, Tyldsley A, Grice EA. Longitudinal Study of the Psoriasis-Associated Skin Microbiome during Therapy with Ustekinumab in a Randomized Phase 3b Clinical Trial. J Invest Dermatol. 2018 Sep;138(9):1973-1981. doi: 10.1016/j.jid.2018.03.1501. Epub 2018 Mar 17. PMID 29559344
- [Derived] Blauvelt A, Ferris LK, Yamauchi PS, Qureshi A, Leonardi CL, Farahi K, Fakharzadeh S, Hsu MC, Li S, Chevrier M, Smith K, Goyal K, Chen Y, Munoz-Elias EJ, Callis Duffin K. Extension of ustekinumab maintenance dosing interval in moderate-to-severe psoriasis: results of a phase IIIb, randomized, double-blinded, active-controlled, multicentre study (PSTELLAR). Br J Dermatol. 2017 Dec;177(6):1552-1561. doi: 10.1111/bjd.15722. Epub 2017 Nov 16. PMID 28600818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During this study, two subjects were transferred between sites and counted twice. Hence, a total of 478 subjects were enrolled in this trial.
Groups:
- Ustekinumab 45 mg/Ustekinumab 90 mg: Open-label period (Week 0-28) - ustekinumab subcutaneous (SC) injections of 45 milligram (mg) at Week 0, 4 and 16 for participants with weight less than or equal to (<=) 100 kilograms (kg) at Week 0 or 90 mg at Week 0, 4, and 16 for participants with weight greater than (>) 100 kg at Week 0.
- Group 1: Approved q12w Maintenance Regimen: Randomized double-blind period (Week 28-124) - Participants who weighed <= 100 kg received 1 ustekinumab SC injection of 45 mg or placebo and participants who weighed > 100 kg received 2 SC injections of ustekinumab 45 mg or placebo.
- Group 2: Subject-tailored Fixed-interval Maintenance Regimen: Randomized double-blind period (Week 28-124) - Participants did not receive a dose of ustekinumab at Week 28. Individual subject-tailored fixed-interval maintenance regimens were determined by observing physician global assessment (PGA) responses from Week 32 through Week 40. The interval separating maintenance doses for each participant was determined by time to loss of PGA response (defined as PGA score of greater than or equal to [>=2]). Participants who weighed <= 100 kg received 1 ustekinumab SC of 45 mg or placebo and participants who weighed > 100 kg received 2 SC injections of ustekinumab 45 mg or placebo.
Period: Open-Label
Arm/Group | Ustekinumab 45 mg/Ustekinumab 90 mg | Group 1: Approved q12w Maintenance Regimen | Group 2: Subject-tailored Fixed-interval Maintenance Regimen
Started | 478 | 0 | 0
Completed | 378 | 0 | 0
Not Completed | 100 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Not all 3 study drug injections received | 2 | 0 | 0
Not completed — Static PGA-cleared/minimal not achieved | 58 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Double-Blind
Arm/Group | Ustekinumab 45 mg/Ustekinumab 90 mg | Group 1: Approved q12w Maintenance Regimen | Group 2: Subject-tailored Fixed-interval Maintenance Regimen
Started | 0 | 76 | 302
Completed | 0 | 59 | 235
Not Completed | 0 | 17 | 67
Not completed — Lost to Follow-up | 0 | 6 | 12
Not completed — Withdrawal by Subject | 0 | 2 | 15
Not completed — Adverse Event | 0 | 4 | 15
Not completed — Death | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 8
Not completed — Protocol Violation | 0 | 0 | 4
Not completed — Pregnancy | 0 | 0 | 3
Not completed — Other | 0 | 2 | 10

BASELINE CHARACTERISTICS:
Population: The "enrolled subject data set" was defined as all participants enrolled at Week 0 who received at least 1 dose of ustekinumab during the study.
Arm/Group | Ustekinumab 45 mg/Ustekinumab 90 mg
Number analyzed (Participants) | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (14.19)
Gender [Count of Participants; unit: Participants]
  Female | 177
  Male | 301
Region of Enrollment [Number; unit: participants]
  United States | 478

OUTCOME MEASURES:

1. Primary Outcome: The Number of Visits at Which Participants Achieved a Static Physician Global Assessment (PGA) Score of Cleared (0) or Minimal (1)
Description: Clinical responses for week (wk)28 sPGA responders randomized to every 12 weeks (q12wk) fixed-interval dosing (Group 1) vs. patient-tailored fixed-interval dosing (Group 2) were assessed using the static PGA (sPGA) measure. Investigators graded psoriasis lesions for induration (0=no plaque elevation to 5=severe plaque elevation), erythema (0=no evidence of erythema to 5=dusky to deep red coloration), and scaling (0=no evidence of scaling to 5=severe scaling). The sum of the 3 scales is divided by 3 and rounded to obtain a final sPGA score, defined as 0=cleared (except for residual discoloration), 1=minimal, 2=mild, 3=moderate, 4=marked or 5=severe.
Time Frame: Up to 24 weeks (Week 88 up to Week 112 [total 7 visits])
Population: The "subjects randomized at Week 28 data set" was defined as the population of enrolled participants who were randomized to either Group 1 or Group 2 at Week 28.
Measure: Mean (95% Confidence Interval); unit: number of visits
Groups:
- Group 1: Ustekinumab q12w Maintenance Regimen (MR): Randomized double-blind period (Week 28-124) - Participants who weighed less than or equal to (<=) 100 kilograms (kg) received 1 ustekinumab subcutaneous injection of 45 milligram (mg) or placebo and participants who weighed > 100 kg received 2 subcutaneous injections of ustekinumab 45 mg or placebo.
- Group 2: Ustekinumab Subject-tailored Fixed-interval MR: Randomized double-blind period (Week 28-124) - Participants did not receive a dose of ustekinumab at Week 28. Individual subject-tailored fixed-interval maintenance regimens were determined by observing physician global assessment (PGA) responses from Week 32 through Week 40. The interval separating maintenance doses for each participant was determined by time to loss of PGA response (defined as PGA score of greater than or equal to [>=2]). Participants who weighed less than or equal to (<=) 100 kilograms (kg) received 1 ustekinumab subcutaneous injection (sc) of 45 mg or placebo and participants who weighed > 100 kg received 2 sc injections of ustekinumab 45 mg or placebo.
Arm/Group | Group 1: Ustekinumab q12w Maintenance Regimen (MR) | Group 2: Ustekinumab Subject-tailored Fixed-interval MR
Number analyzed (Participants) | 76 | 302
number of visits | 4.5 (3.07) [3.81 to 5.21] | 4.1 (2.93) [3.72 to 4.39]

2. Secondary Outcome: The Percentage of Participants With a Static PGA Score of Cleared (0) or Minimal (1) Over Time
Description: Clinical responses for week (wk) 28 sPGA responders randomized to every 12 weeks (q12wk) fixed-interval dosing (Group 1) vs. patient-tailored fixed-interval dosing (Group 2) were assessed using the static PGA (sPGA) measure. Investigators graded psoriasis lesions for induration (0=no plaque elevation to 5=severe plaque elevation), erythema (0=no evidence of erythema to 5=dusky to deep red coloration), and scaling (0=no evidence of scaling to 5=severe scaling). The sum of the 3 scales is divided by 3 and rounded to obtain a final sPGA score, defined as 0=cleared (except for residual discoloration), 1=minimal, 2=mild, 3=moderate, 4=marked or 5=severe.
Time Frame: Week 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112
Population: The Analysis population was "subjects randomized at Week 28 data set". 'n' signifies number of participants who were evaluable at each specific timepoint, for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Ustekinumab q12w Maintenance Regimen (MR) | Group 2: Ustekinumab Subject-tailored Fixed-interval MR
Number analyzed (Participants) | 76 | 302
percentage of participants
  Week 28 (n=76, 302) | 100 | 100
  Week 32 (n=75, 297) | 78.7 | 71.0
  Week 36 (n=74, 288) | 75.7 | 59.0
  Week 40 (n=73, 280) | 67.1 | 56.4
  Week 44 (n=71, 278) | 74.6 | 68.3
  Week 48 (n=69, 269) | 69.6 | 69.9
  Week 52 (n=69, 274) | 71.0 | 66.4
  Week 56 (n=68, 271) | 73.5 | 61.3
  Week 60 (n=68, 268) | 70.6 | 67.9
  Week 64 (n=69, 268) | 59.4 | 65.7
  Week 68 (n=69, 264) | 75.4 | 57.2
  Week 72 (n=66, 262) | 74.2 | 63.7
  Week 76 (n=66, 264) | 60.6 | 58.7
  Week 80 (n=65, 258) | 67.7 | 53.5
  Week 84 (n=63, 258) | 68.3 | 55.0
  Week 88 (n=64, 257) | 57.8 | 60.7
  Week 92 (n=64, 254) | 65.6 | 57.9
  Week 96 (n=62, 254) | 58.1 | 56.3
  Week 100 (n=64, 250) | 59.4 | 50.8
  Week 104 (n=65, 250) | 64.6 | 56.4
  Week 108 (n=63, 244) | 60.3 | 58.6
  Week 112 (n=58, 242) | 53.4 | 55.0

3. Secondary Outcome: The Number of Visits for Which Participants Achieved a Psoriasis Area and Severity Index (PASI) 75 Response
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 to 72. A PASI 75 response is defined as greater than or equal to (>=) 75 percent (%) improvement in PASI score from baseline.
Time Frame: Up to 24 weeks (Week 88 up to Week 112 [total 7 visits])
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Group 1: Ustekinumab q12w Maintenance Regimen (MR) | Group 2: Ustekinumab Subject-tailored Fixed-interval MR
Number analyzed (Participants) | 76 | 302
number of visits | 5.8 (2.31) | 5.4 (2.61)

4. Secondary Outcome: The Percentage of Participants With a PASI 75 Response Over Time
Description: as for outcome 3
Time Frame: Week 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, 104, 108, 112
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Group 1: Ustekinumab q12w Maintenance Regimen (MR) | Group 2: Ustekinumab Subject-tailored Fixed-interval MR
Number analyzed (Participants) | 76 | 302
percentage of participants
  Week 28 (n=76, 302) | 96.1 | 95.7
  Week 32 (n=75, 297) | 92.0 | 81.1
  Week 36 (n=74, 288) | 93.2 | 78.8
  Week 40 (n=73, 280) | 86.3 | 77.5
  Week 44 (n=71, 278) | 90.1 | 83.5
  Week 48 (n=69, 269) | 89.9 | 82.9
  Week 52 (n=69, 274) | 82.6 | 84.7
  Week 56 (n=68, 271) | 85.3 | 83.8
  Week 60 (n=68, 268) | 91.2 | 82.8
  Week 64 (n=69, 268) | 79.7 | 83.2
  Week 68 (n=69, 264) | 85.5 | 79.9
  Week 72 (n=66, 262) | 83.3 | 83.6
  Week 76 (n=66, 264) | 77.3 | 79.9
  Week 80 (n=65, 258) | 81.5 | 76.4
  Week 84 (n=63, 258) | 84.1 | 74.8
  Week 88 (n=64, 257) | 81.3 | 78.2
  Week 92 (n=64, 254) | 84.4 | 77.2
  Week 96 (n=62, 254) | 82.3 | 79.1
  Week 100 (n=64, 250) | 76.6 | 75.6
  Week 104 (n=65, 250) | 81.5 | 79.2
  Week 108 (n=63, 244) | 82.5 | 79.9
  Week 112 (n=58, 242) | 74.1 | 77.7

ADVERSE EVENTS:
Time Frame: Week 0 through Week 124
Description: During this study, 5 pregnancies were reported in female participants in Group 2, and 2 pregnancies were reported in partners of male participants in Group 2.
Arm/Group | Ustekinumab 45 mg/Ustekinumab 90 mg | Group 1: Approved q12w Maintenance Regimen | Group 2: Subject-tailored Fixed-interval Maintenance Regimen
Serious Adverse Events (participants affected / at risk) | 14/478 | 7/76 | 21/302
Other Adverse Events (participants affected / at risk) | 73/478 | 39/76 | 131/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab 45 mg/Ustekinumab 90 mg (N=478) | Group 1: Approved q12w Maintenance Regimen (N=76) | Group 2: Subject-tailored Fixed-interval Maintenance Regimen (N=302)
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 — During this study, a total of 2 deaths were reported. 1 participant in Group 1 died of natural causes and reported as an SAE of Death, and 1 participant in Group 2 died as an outcome of Acute Myeloid Leukemia (AML) and reported as an SAE of AML.
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Abscess Limb (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Appendicitis Perforated (Infections and infestations) | 1 | 0 | 0
Bacterial Infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Carotid Artery Occlusion (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Drug Withdrawal Convulsions (Nervous system disorders) | 1 | 0 | 0
Viith Nerve Paralysis (Nervous system disorders) | 1 | 0 | 0
Homicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 1 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hernia Diaphragmatic Repair (Surgical and medical procedures) | 1 | 0 | 0
Knee Arthroplasty (Surgical and medical procedures) | 0 | 1 | 0
Spinal Laminectomy (Surgical and medical procedures) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ustekinumab 45 mg/Ustekinumab 90 mg (N=478) | Group 1: Approved q12w Maintenance Regimen (N=76) | Group 2: Subject-tailored Fixed-interval Maintenance Regimen (N=302)
Nasopharyngitis (Infections and infestations) | 24 | 7 | 47
Sinusitis (Infections and infestations) | 6 | 3 | 17
Upper Respiratory Tract Infection (Infections and infestations) | 25 | 21 | 59
Urinary Tract Infection (Infections and infestations) | 7 | 4 | 9
Transaminases Increased (Investigations) | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 16
Hypertension (Vascular disorders) | 4 | 6 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.